CLINICAL TRIAL: NCT06130995
Title: Phase IB Trial of Relugolix and Enzalutamide as Neoadjuvant/ Adjuvant to Local-regional Treatment in Patients With High-risk Locally Advanced Prostate CAncer (RENAPCA)
Brief Title: Relugolix + Enzalutamide Study in High-Risk Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Pfizer (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-RENAPCA
Record Dates: First submitted 2023-11-07; First posted 2023-11-14 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Androgen Deprivation Therapy; Locally Advanced Prostate Cancer
Keywords: dose limiting toxicity (DLTs); pathologic complete response (pCR); minimal residual disease (MRD); radiation therapy (RT)
MeSH Terms: conditions — Pathologic Complete Response; Neoplasm, Residual | interventions — relugolix; enzalutamide

STUDY DESIGN:
Intervention Model Description: This is a single arm phase Ib study with safety lead-in cohorts to investigate the efficacy and safety of neoadjuvant and adjuvant hormonal therapy with relugolix plus enzalutamide in patients with high-risk locally advanced prostate cancer who are candidates for ADT followed by definitive radiation therapy (RT) or surgical treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate Cancer Combo Therapy Trial (Experimental): A single-arm Phase Ib study explores the effectiveness and safety of neoadjuvant and adjuvant hormonal therapy combining relugolix and enzalutamide in high-risk locally advanced prostate cancer patients eligible for ADT followed by radiation therapy or surgery.
  Interventions: Drug: Relugolix and Enzalutamide

INTERVENTIONS:
Drug: Relugolix and Enzalutamide — Dose level of Relugolix and Enzalutamide Safety Lead-in Cohort, 3-12 patient. Relugolix;120 mg, oral, once daily, with a loading dose of 360 mg on day 1, Enzalutamide; 120-160 mg, oral, once daily.
  Dose Expansion Cohort, up to 34 patients. Relugolix;120 mg, oral, once daily, with a loading dose of 360 mg on day 1, Enzalutamide; To be determined by safety lead-in cohort.
  One cycle = 3 months The dose limiting toxicity (DLT) period is the first 28 days
  Neoadjuvant ADT: 6 months; Relugolix: 120 mg orally, daily (with a 360 mg loading dose on day 1, Enzalutamide: 160 mg (or 120 mg) orally, daily
  Concurrent ADT during Radiation Therapy; Relugolix: 120 mg orally, daily (with a 360 mg loading dose on day 1, Enzalutamide: 160 mg (or 120 mg) orally, daily
  Maintenance ADT: Additional 18 months; Relugolix: 120 mg orally, daily (with a 360 mg loading dose on day 1, Enzalutamide: 160 mg (or 120 mg) orally, daily

SUMMARY:
The goal of this clinical trial is to test how effective and safe it is to use a combination of two medications, relugolix and enzalutamide, in patients with advanced prostate cancer. We want to see if this combination can help improve the chances of curing the cancer and make the patients live longer without the cancer getting worse.

The main questions we want to answer in this study are:

* Can using relugolix and enzalutamide together help increase the chances of curing high-risk advanced prostate cancer?
* Does this combination treatment help patients live longer without their cancer getting worse?

Participants in this study will be asked to take relugolix and enzalutamide as part of their cancer treatment. They will also undergo Radiation Therapy or prostatectomy, which are standard treatments for this type of cancer.

DETAILED DESCRIPTION:
This clinical trial aims to assess the effectiveness and safety of combining relugolix and enzalutamide as neoadjuvant and adjuvant androgen deprivation therapy (ADT) in patients diagnosed with high-risk locally advanced prostate cancer who are also candidates for definitive radiation therapy (RT) or surgical treatment. The objectives of this phase Ib clinical trial are to evaluate the efficacy, safety, and dynamic changes in biomarkers associated with this combination therapy. A combined total of up to 41 evaluable patients will participate in this study, with the initial safety lead-in cohorts involving a potential enrollment of 12 patients, followed by a dose expansion cohort that may include up to 29 subjects.

The combined treatment cycle spans 28 days, with patients receiving six months of neoadjuvant therapy followed by an additional 18 months in the adjuvant setting. Treatment duration may be shortened if unacceptable toxicity occurs or if a patient withdraws consent. Approximately 24 months of post-accrual follow-up are anticipated to adequately assess the efficacy and safety of the treatment.

Ultimately, the study aims to contribute valuable insights into the potential benefits of neoadjuvant and adjuvant hormonal therapy with relugolix plus enzalutamide in improving outcomes for patients facing high-risk locally advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent;
2. Patients must be ≥18 years of age at the time of signing the informed consent form.
3. Men with a diagnosis of adenocarcinoma of the prostate pathologically proven diagnosis with the following:

   • Locally advanced high-risk prostate defined as i. PSA >20 ng/mL or ISUP grade 4/5 (Gleason score >7) or cT2c or ii. Any PSA, any ISUP grade, cT3-4 or cN+ (locally advanced)
4. Have normal organ and bone marrow function measured at the screening visit including

   * Platelets ≥100 × 103/microliter (μL);
   * Hemoglobin ≥ 10.0 grams/dL;
   * Leukocytes (WBC) ≥ 3 × 103/μL;
   * Absolute neutrophil count ≥1.5 × 103/μL;
   * Serum AST and ALT ≤2.5 × upper limit of normal (ULN);
   * Total bilirubin ≤1.5 ×ULN (unless values are consistent with Gilbert's syndrome for which the total bilirubin must be < 3x ULN);
   * Serum creatinine ≤ 1.5 × ULN; OR Measured or calculated creatinine clearance ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
6. The participant has, in the opinion of the investigator, a life expectancy of at least 6 months.
7. Male patients must be willing to use contraception during treatment and for 3 months after the last dose of study treatment when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential.

Exclusion Criteria:

1. History of major adverse cardiac event, including myocardial infarction, new congestive heart failure (CHF) or CHF exacerbation, or stroke, within the past 6 months.
2. Patients who are receiving any other investigational agents.
3. Patients with distant metastatic cancer will be excluded from the study as intermittent hormonal therapy is not standard of care treatment for this population.
4. Active secondary malignancies requiring treatment
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to any of study drugs
6. Participants with uncontrolled intercurrent illness.
7. Participant is unable to swallow pills.
8. Not a candidate for surgical or radiation therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient experiencing dose limiting toxicity (DLT) and tolerable dose of relugolix and enzalutamide combination | 2-3 years
  Proportion of patients will undergo evaluation for dose-limiting toxicity (DLT) to establish a tolerable dosage regimen for the combined use of relugolix and enzalutamide in individuals diagnosed with high-risk locally advanced prostate cancer. The assessment hinges on identifying DLTs associated with this treatment using 3-12 patients from the safety lead-in cohort and continuously monitoring treatment-related adverse events throughout the DLT observation period, which spans 24 months, encompassing neoadjuvant and adjuvant treatment phases.
Proportion of patients experiencing Pathologic Complete Response (pCR) and Minimal Residual Disease (MRD) in Neoadjuvant ADT with the combination of Relugolix and Enzalutamide | 4-6 years
  Proportion of patients achieving a pathologic response rate, defined as the combined Pathologic Complete Response (pCR) Rate and Minimal Residual Disease (MRD) rate (MRD, tumor ≤5 mm), serves as the primary endpoint for the dose expansion cohort. This assessment will be conducted using Simon's optimal 2-stage design, enabling a determination of whether there are an adequate number of patients with objective responses to proceed to the second stage of the study (at the interim analysis) or to consider the drug for further investigation in a Phase III study (at the study's conclusion).

SECONDARY OUTCOMES:
Objective response rate (ORR) of neoadjuvant ADT of relugolix and enzalutamide | 4-6 years
  Assessing the objective response rate (ORR) in patients with high-risk locally advanced prostate cancer eligible for definitive radiation therapy (RT) or radical prostatectomy, following neoadjuvant ADT with relugolix and enzalutamide. ORR will be determined based on MRI imaging confirmation, defined as the percentage of patients achieving a complete response (CR) or partial response (PR) per RECIST v1.1 criteria.
Frequency and severity of adverse events of relugolix and enzalutamide | 4 years
  Assessment includes the rate and severity of treatment-related adverse events as per the NCI CTCAE v5 grading system.
Prostate specific antigen (PSA) response to the combination of relugolix and enzalutamide | 4 years
  Measurement of prostate-specific antigen (PSA) response, includes the rate and duration of a 50% reduction in PSA levels from baseline.
Diagnostic precision and constraints of biopsy in assessing positive margin rates and rates of pathologic downgrade. | 4-6 years
  Assessments involves diagnostic capabilities of biopsy-based analysis for prostatectomy, as reflected in the rates of positive margin in whole-mount pathology following intense neoadjuvant therapy and the pathologic downgrade compared to the initial T stage.
Progression-Free Survival (PFS) in Patients Receiving Neoadjuvant Relugolix and Enzalutamide | 4-6 years
  Assessment of Progression-Free Survival (PFS); defined as the interval from the initial dose to the earliest evaluation of progression according to RECIST v1.1 criteria, in patients undergoing neoadjuvant treatment with Relugolix and Enzalutamide, followed by radical local-regional Radiation Therapy (RT) or Radical Prostatectomy (RP) and subsequent adjuvant maintenance Androgen Deprivation Therapy (ADT).

CONTACTS AND LOCATIONS:
Locations (1):
- Stephenson Cancer Center at OU Health, University of Oklahoma Health Sciences Center (SCC-OUHSC), Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No